CLINICAL TRIAL: NCT01301794
Title: Study of the Effects of Lovaza (Omega 3 Fatty Acids) On Lipoprotein Particles and Their Transcriptional Effects
Brief Title: Lovaza Mechanisms of Action
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Jorge Plutzky, Director of Vascular Disease Prevention Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BWHp001640
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Moderate Hypertriglyceridemia.
Keywords: Hypertriglyceridemia; Fish oil; Omega 3 fatty acids
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Fatty Acids, Omega-3; Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Omega 3 fatty acid (Lovaza) — Lovaza is an FDA approved omega 3 fatty acid taken as 4 grams a day (two one gram formulations twice a day).
  Other Names: Lovaza LVZ112737, formerly known as Omacor.; Omega 3 fatty acids are also available over the counter but Lovaza is a proprietary form.

SUMMARY:
High levels of triglycerides is a common abnormality found in patients with diabetes and also cardiovascular disease, and may contribute to the risk for both. Omega 3 fatty acids, as found enriched in fish and also in the commercial agent called Lovaza lower triglyceride levels. Prior work from the investigators group demonstrated that an enzyme responsible for the break down of triglycerides - lipoprotein lipase - generates molecules that can activate a specific nuclear receptor known as PPAR-alpha. This study investigates the hypothesis that taking Lovaza shifts the specific fatty acid content of triglyceride containing lipoproteins and increases the ability of those lipoproteins to activate PPAR-alpha.

DETAILED DESCRIPTION:
This study will investigate changes in lipid and other metabolic parameters as well as the ability of isolated lipoproteins to activate PPARs in the presence or absence of lipoprotein lipase in a cohort of normal healthy individuals with modest hypertriglyceridemia before and after a course of Lovaza.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy 21 to 65 year old men and women
* Triglycerides >150 < 500 mg/dL

Exclusion Criteria:

* Other lipid lowering medication including fish oil
* Major illnesses
* Diabetes
* Cardiovascular disease
* Abnormalities uncovered on screening blood work including undiagnosed diabetes, abnormal liver function tests, triglycerides > 500 mg/dL
* Indication for immediate statin therapy
* Pregnancy
* Contraindication for fish oil use or muscle biopsy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Changes in lipoprotein metabolite content and their ability to activate PPAR-alpha in an established cell culture system. | 3 months
  Enrolled subjects will serve as their own controls and will be studied at baseline and after 3 months of Lovaza. The primary endpoint will test changes in lipoproteins as a function of their content and ability to activate PPAR-alpha in standard transfected cell culture systems.

SECONDARY OUTCOMES:
Changes in plasma markers for atherosclerosis | 3 months
  Subjects will also be studied before and after Lovaza for changes in lipid profile and c- reactive protein
Change in plasma markers of diabetes | 3 months
  Plasma markers of diabetes will be measure before and after Lovaza treatment for 3 months, specifically glucose and A1C levels
Changes in plasma markers of liver function | 3 months
  Plasma levels of liver function tests, specifically ALT and AST before and after 3 months of Lovaza.
  This is not a safety issue since elevated triglycerides can cause increased liver function tests and fish oil (like Lovaza) can lower triglyceride levels and hence ALT and AST levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Plutzky, MD, Principal Investigator — Brigham and Women's Hospital; Jonathan Brown, MD, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States